CLINICAL TRIAL: NCT04688463
Title: Evaluation of Pressure Algometry in the Clinical Assessment of Acute Abdominal Pain in Children
Status: Completed | Type: Observational
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Ray Postuma, Professor of Surgery - retired, University of Manitoba
Other Study IDs: H2003:104
Record Dates: First submitted 2020-12-21; First posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Appendicitis; Diagnoses Disease; Pediatric ALL
Keywords: Appendicitis; Children; Diagnosis; Pressure-Pain Algometry
MeSH Terms: conditions — Appendicitis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this retrospective observational case study, the investigators review the clinical experience with pressure-pain algometry in children with suspected appendicitis. The investigators hypothesized that algometry can discriminate children with appendicitis from children without appendicitis and aimed to determine the diagnostic accuracy of algometry, compared to ultrasound imaging and clinical assessment.

DETAILED DESCRIPTION:
As a retrospective cohort study, participants include all children referred with abdominal pain from January 2000 to June 2006 to one surgeon (R.P.) on the pediatric general surgery service at the Health Sciences Centre (HSC)-Children's Hospital in Winnipeg. The HSC-Children's Hospital is the only pediatric surgery centre within a radius of 600 km. All included participants have had acute abdominal pain ≤ 7 days, and suspected appendicitis based on standard history and physical exam. Standard appendicitis treatments were used: analgesia, antibiotics, operation. The Research Ethics Board of the University of Manitoba approved the study and reporting of the findings (H2003:104).

The investigators use standard clinical, laboratory, diagnostic imaging procedures for appendicitis diagnosis. The final diagnosis is defined by:

* pathology report indicating transmural inflammation, or
* from the surgeon's report when pathology was unavailable, or
* by discharge diagnosis in non-operated patients.

Appendix rupture is defined by the presence of pus and full-thickness perforation of the appendix wall or abscess formation at operation or on pathology examination. The appendix condition is classified as normal, non-perforated or perforated; all other pathologies at operation are recorded. Treatments, complications and morbidity are tabulated.

Clinical Measures

All patient demographics, clinical presentation details, and results of laboratory testing (WBC) are collated. From this, the components of the Alvarado and Samuel pediatric appendicitis scores (PAS) are calculated retrospectively for comparison purposes and not used in patient management. Time intervals are calculated from the date and time entries in the clinical record. Results of diagnostic abdominal imaging (U/S, CT, plain x-rays) are based on recorded verbal or, if available, official written reports at the time of patient management decision. Equivocal imaging results are deemed negative. The reasons why algometry was not done are tabulated and the number of patients who reached or exceeded the maximum algometer readout (≥4 kg)

Algometry Device and Procedure:

The principal investigator (PI) designed and produced in 1983 a simple, lightweight, aluminum-Teflon®, pocket-size, calibrated spring-gauge algometer, similar to a tire gauge, that was used for all measurements. The PI used this routinely in his clinical work.

Children were first familiarized with the algometer and allowed to hold and play with it. The device head was then depressed with increasing force to the child's unencumbered mid-forearm to simulate the abdominal examination and algometry procedure. Children were instructed to indicate with their preferred 'signal' (e.g. 'now', 'ow!', or squeezing the examiner's fingers) when the sensation of pressure changed to a sensation of discomfort or pain. Pressure-pain threshold (PPT) is defined as the minimum force (in kilograms) applied via the algometer to produce discomfort. Lower PPT readings imply greater tenderness. All measurements were obtained and recorded by the Principal Investigator. Algometry was a standard tool used by the PI in all clinical practice.

Single mid-forearm 'pressure-pain threshold algometry' (PPTA) measurements are used as the patient's background, 'global', non-abdominal discomfort/pain threshold. This was then followed by single PPTA measurements from the centre of each four abdominal quadrants in the following sequence: left lower quadrant, left upper quadrant, right upper quadrant and right lower quadrant. The lower quadrant centre was defined midway between the umbilicus and anterior iliac spines. The upper quadrant centre was defined midway between the umbilicus and mid-costal margins. Algometer depressing velocity (rate) mimicked normal, heuristic palpation velocity (i.e. approximately 1 kg./sec (0.241 kg/cm2/sec or 23.6 kilopascal/sec). From the 5 sites, the investigators define 7 pressure-pain threshold algometric measurements of interest (forearm, left lower quadrant, left upper quadrant, right upper quadrant and right lower quadrant, lowest reading, average reading).

Additional algometry 'mapping' is done when the most tender site apparent on qualitative palpation was outside the standard four abdominal quadrants e.g. suprapubic or flank tenderness. If the algometry measurements and qualitative assessment agreed, patients are classified as 'concordant' versus 'discordant' when no agreement. For purposes of analysis, 'discordant' patients are included with the non-mapped group. The site of these maximal abdominal wall tenderness measurements are then correlated with the location of the inflamed appendix found at operation.

The primary analysis is with baseline algometry readings or the final of serial readings. The algometry readings of non-appendicitis appendectomy patients are grouped with non-appendicitis patients.

When available and appropriate, algometry measures are repeated during the period of diagnostic observation to determine if serial PPTA 'mirrored' the patient's clinical course.

From these algometry measures the following ratios are determined:

* Abdominal tenderness localizing ratio (ATLR), calculated as the ratio of abdominal tenderness between the least tender (highest PPT) and most tender (or RLQ) quadrants. A higher ATLR indicates a greater degree of tenderness localization within the abdomen; lower ATLR indicates more diffuse tenderness.
* Global abdominal tenderness localizing ratio (GTLR), calculated as the ratio of the forearm and most tender (or RLQ) quadrant's (lowest PPT) reading. Higher GTLR indicates a greater degree of tenderness localized to the abdomen relative to the patient's global discomfort/pain threshold. Patients thus serve as their own tenderness control.

For analysis of correlation with clinical variables, the Pearson correlation coefficient R2, are calculated between the 7 PPTA's and age, weight (expressed as a percentile), and duration of symptoms, stratified by gender.

To assess the discriminatory power and predictive values of algometry, we randomly split the data into derivation and validation groups, stratify to gender and final diagnosis of appendicitis. Receiver operating characteristic (ROC) analysis is then performed to identify the area under the curve (AUC), sensitivity, specificity, positive and negative predictive values (PPV and NPV) of algometry. The diagnostic accuracy of algometry is compared to ultrasound assessment and clinical diagnosis, again stratified to gender. GraphPad™ is used for all the statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* all children referred with abdominal pain from January 2000 to June 2006 to one surgeon on the pediatric general surgery service at the Health Sciences Centre (HSC)-Children's Hospital in Winnipeg.

Exclusion Criteria:

* children with abdominal pain > 7 days
* children with abdominal pain due to other surgical or medical conditions

Ages: 2 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: -included participants have had acute abdominal pain ≤ 7 days, and suspected appendicitis based on standard history and physical exam; consecutive participant sampling
Sampling Method: Probability Sample
Enrollment: 427 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2006-06-15 (Actual); Study Completion 2006-06-15 (Actual)

PRIMARY OUTCOMES:
Appendicitis | within 1 week
  Diagnosis of appendicitis as confirmed at operation
Appendicitis | within 1week
  Diagnosis of appendicitis by pathology report if available.
Non-Appendicitis | Within one (1) week
  Diagnosis of non-appendicitis by observation only
Pressure-pain algometry | Within one (1) week
  Single measurements taken before final management decision
Pressure-pain algometry | Within one (1) week
  Serial measurements taken before final management decision

SECONDARY OUTCOMES:
Complications following appendectomy | For one (1) month following operation or observation.
  Categorization of all postoperative complication including deaths